## INFORMED CONSENT OF THE PATIENT'S LEGAL GUARDIAN TO PARTICIPATE IN THE RESEARCH STUDY

| Assessment of motor skills, incidence of musculoskeletal injuries, quality of life and nutrition among children and adolescents participating in sport as part of the Healthy Sport for Children and Adolescents Project |
|---|
| I, the undersigned(s), declare that I have read and understood the above information regarding the described clinical trial and have received comprehensive answers to my satisfaction to the questions asked. I voluntarily consent to the participation of my child |
| I have been informed that the data controller will be the facility where the study is being carried out, that I have the right to inspect and correct my child's data and that the data is provided voluntarily. By signing this document, I also confirm that I have been informed about how the data from the study will be processed and that the data will be verified by comparing them with my child's medical records, and that the data are only collected for the scientific analysis of the study. |
| I consent to the processing of my child's data in this study in accordance with the laws in force in Poland (Personal Data Protection Act of 29.08.1997). I consent to the transfer of my child's anonymised data to other countries, both within and outside Europe. The data analysed by the investigators and the Bioethics Committee will only be available in anonymous form. I have been informed that if I withdraw my consent for my child to participate in the study, the data collected so far may be used and processed as part of the study database. |
| I consent to photographs being taken of my child for the purpose of movement analysis for the study. |
| Consent is drawn up in duplicate. |
| Patient's legal guardian: |
| Name Signature Date of signature (in block capitals) |
| I declare that I have discussed the study presented with the parent/legal guardian of the patient/patient using clear wording that is as simple as possible and have provided information on the nature and significance of the study. |
| Consenting person |
| WILCZYŃSKI BARTOSZ |

Informed consent form version 1 dated 15.01.2023

Name (in block capitals) Signature Date of signature